CLINICAL TRIAL: NCT03525821
Title: Intranasal Ketamine Use in the Management of Upper Limb's Fracture Reduction in Pediatric Emergencies
Brief Title: Intranasal Ketamine and Fracture Reduction in Pediatric Emergencies (KETAPED)
Acronym: KETAPED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-HPNCL-01
Record Dates: First submitted 2018-04-20; First posted 2018-05-16 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Fractures, Closed
MeSH Terms: conditions — Fractures, Closed | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intranasal administration of ketamine (Experimental): intranasal adminstration of ketamine combined with nitrous oxide befor reduction of fracture
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — intranasal use of ketamine 1mg/kg with nitrous oxide

SUMMARY:
The incidence of child fractures is around 180 per 10,000 children under 16 years old in industrialized countries. More and more hospitals, such as Nice University Hospital, are using vigilant procedural sedation for simple surgical procedures such as fracture reduction, allowing ambulatory care. This is why the investigators propose the alternative of intranasal ketamine associated with nitrous oxide inhalation in the management of children's pain. Indeed, thanks to its short duration of action and short duration of effectiveness, ketamine is already used in pediatric anesthesia and resuscitation for many years and is considered safe and effective.

The objective of this work is to evaluate the efficacy of intranasal ketamine associated with nitrous oxide inhalation in the reduction of isolated fractures from the extremity of the upper limb in children allowing optimal management.

This work will consist of research involving non-randomized, monocentric prospective interventional category 1 for duration of 18 months. Patients over 4 years of age and under 18 years, with a closed fracture isolated from the distal extremity of the upper limb, with stable hemodynamic will be included. In view of active queue of pediatric emergencies Nice University Hospital, the investigators can include 60 patients, allowing to have a representative sample of the pediatric population.

The treatment administered will be intranasal ketamine, using a tip MAD® (Mucosal Atomization Device) at a dosage of 1 mg/kg in a single administration, under continuous cardiorespiratory monitoring for 2 hours. The reduction of the fracture will be done under inhalation of nitrous oxide. The primary endpoint will be pain control during and after fracture reduction, defined by the FLACC Hetero-Assessment Pain Rating Scale. Others parameters as the evaluation of the degree of sedation, evaluation of the child's feeling of pain after the reduction, evaluation of the feasibility of the preparation and administration of the drug by the nurse will be reported.

DETAILED DESCRIPTION:
The incidence of child fractures is around 180 per 10,000 children under 16 years old in industrialized countries (Norway, Sweden, Great Britain and France). However, the rate of fractures treated in pediatric emergencies varies according to the different sports activities and the location of the hospital. In Nice, the number of fractures of the upper limb in children is about 400 per year, because of the sporting diversity between sea and mountains to which children have access.

Most of the child's fractures are treated in operating theaters in hospitals in France. However, more and more hospitals, such as Nice University Hospital, are using vigilant procedural sedation for simple surgical procedures such as fracture reduction, allowing ambulatory care. At the University Hospital of Nice, analgesic management of simple fractures of the child, including fractures of the upper limb, combines 2 drugs: midazolam and nalbuphine intra-rectal. This therapy is used in combination with nitrous oxide inhalation for the reduction of the fracture site.

However, this treatment is not optimal: midazolam has significant side effects (respiratory depressant, hypotensive, excessive drowsiness, etc.) and the intrarectal way of administration suggests a problem of delayed action of the administered product, causing a variability of the effectiveness of the drug over time and a social problem. This is why the investigators propose the alternative of intranasal ketamine associated with nitrous oxide inhalation in the management of children's pain. Indeed, thanks to its short duration of action and short duration of effectiveness, ketamine is already used in pediatric anesthesia and resuscitation for many years and is considered safe and effective. This drug is a very interesting choice in the treatment of analgesics in surgical emergencies. However, it is not used in pediatric emergencies for excessive fear of side effects and service habits.

The objective of this work is to evaluate the efficacy of intranasal ketamine associated with nitrous oxide inhalation in the reduction of isolated fractures from the extremity of the upper limb in children allowing optimal management.

This work will consist of research involving non-randomized, monocentric prospective interventional category 1 for a duration of 18 months. Patients over 4 years of age and under 18 years, with a closed fracture isolated from the distal extremity of the upper limb, with stable hemodynamic will be included. In view of active queue of pediatric emergencies Nice University Hospital and taking into account lost sight, the investigators can include 60 patients, allowing to have a representative sample of the pediatric population.

The treatment administered will be intranasal ketamine, using a tip MAD® (Mucosal Atomization Device) at a dosage of 1 mg/kg in a single administration, under continuous cardiorespiratory monitoring for 2 hours. The reduction of the fracture will be done under inhalation of nitrous oxide.

The primary endpoint will be pain control during and after fracture reduction, defined by the FLACC Hetero-Assessment Pain Rating Scale < 4/10.

The secondary evaluation criteria will be: the evaluation of the degree of sedation during the gesture by the "University of Michigan Sedation Scale" score, the evaluation of the tolerance of the treatment in the child during and after the gesture (presence of desaturation) O2 <94%, hypersialorrhea, apnea, laryngospasm), evaluation of the child's feeling of pain after the reduction, evaluation of the feasibility of the preparation and administration of the drug by the nurse.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Children
* Aged 4 to 17 years old
* Presenting a fracture isolated from the distal end of the upper limb with closed focus, requiring a reduction
* Fracture dating from <72h
* stable hemodynamics
* Affiliation to a social security scheme
* Signature of the authorization documents of the 2 parents or the representative of the parental authority for the participation of the child in the study
* Signature of informed consent for children over 15 years of age

Exclusion Criteria:

* Known hypersensitivity to ketamine
* History of epilepsy or known psychiatric illness
* Any child with a developing respiratory disease (asthma, laryngitis, tracheitis)
* Any child who has received an analgesic of level 2 or 3 in the 3 hours preceding the treatment in pediatric emergencies
* High Blood Pressure
* Severe Heart Failure
* polytrauma
* Open fracture
* Proven pregnancy
* Any child requiring pure oxygen ventilation.
* Nitrous oxide should not be used in situations at risk of accumulation in cavities and when its expansion could be dangerous, such as cranial trauma with alteration of the state of consciousness, maxillofacial trauma, pneumothorax, gas embolism , bullous emphysema, sinus or middle ear surgery, internal ear surgery, severe abdominal distension (eg, bowel occlusion)
* A child who has recently received an ophthalmic gas (SF6, C3F8, C2F6) used in ocular surgery as long as a gas bubble persists inside the eye and at a minimum for a period of 3 months. Severe post-operative complications may occur in relation to increased intraocular pressure

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-09-13 (Actual); Study Completion 2020-09-13 (Actual)

PRIMARY OUTCOMES:
effectiveness evaluation of ketamine by measure the change of pain control | 5 minutes before the admintration of the ketamine and 15 min and 30 min after the administration of the ketamine
  The effectiveness of ketamine will be assessed by measuring the change of pain control between the baseline and after fracture reduction.
  Measurement of pain intensity will be carried out using the Face, Legs, Activity, Cry, Consolability scale (FLACC) 5-item hetero-evaluation of pain, validated in children. The FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
  Effective pain control will be defined by a score obtained with the FLACC <4/10 scale during reduction and after reduction. Our criterion will therefore be binary: control or not control of pain.

SECONDARY OUTCOMES:
evaluation of the degree of sedation | 5 minutes after the administration of the ketamine
  The evaluation of the degree of sedation will be made 5 minutes after the administration of the ketamine by the internationally validated anesthetic score "University of Michigan Sedation Scale" based on 5 items ranging from the state of awakening to no response to stimulation.
  The level of sedation sought is a score equal to 1 corresponding to a relaxed / sleeping patient and having an appropriate response to the weak stimulation.
evaluation of tolerance | from time of ketamine administration to the end of patient participation of study, for about 3 hours
  Treatment tolerance in children will be assessed through the collection of adverse reactions for the duration of the procedure, from the introduction of sedation to the end of the post-reduction period .
  Possible side effects are listed in "Undesirable Events" section in CRF. For each adverse event, the patient rate with at least one occurrence of the effect should be determined.
evaluation of child's feeling of pain | after the reduction during 2 hours
  The assessment of the child's feeling of pain after the reduction will be carried out by a closed question:
  "Have you had any pain?" Possible answers: No, Yes a little, Yes a lot
The nurse's assessment of preparation feasibility of ketamine | 30 minutes after the preparation of the treatment
  The nurse's assessment of the feasibility of the preparation of the medicinal product will be based on a questionnaire based on two closed questions on the timeliness of drug preparation :
  "Are you satisfied with the speed of preparation of intranasal ketamine? " Answers: Not satisfied, Partially satisfied, Satisfied, Very satisfied
The nurse's assessment of administration feasibility of ketamine | 30 minutes after the administration of the treatment
  The nurse's assessment of the feasibility of the administration of the medicinal product will be based on a questionnaire based on two closed questions on the ease of administration of the drug intranasally: Are you satisfied with the ease of administration of intranasal ketamine? " Answers: Not satisfied, Partially satisfied, Satisfied, Very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure HERISSE, MD, Principal Investigator — Hôpitaux Pédiatriques de Nice CHU-LENVAL
Locations (1):
- Hôpitaux pédiatriques de Nice CHU-Lenval, Nice, France